CLINICAL TRIAL: NCT06437223
Title: A Phase 2 Study to Compare the Efficacy and Safety of Orally Administered Xiflam™ Therapy With Orally Administered Placebo in Patients With Ocular and Systemic Manifestations of Post COVID Sequelae Known as "Long" COVID
Brief Title: Study of Xiflam™ Treatment in Patients Post COVID-19 Infection Suffering From What is Known as Long COVID (LC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inflammx Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFX-LC001
Record Dates: First submitted 2024-05-16; First posted 2024-05-31 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-05

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — tonabersat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 2 randomized, masked, placebo-controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): IFX-LC001 Tonabersat tablets 40mg tablets or placebo Take two tablets once per day
  Interventions: Drug: Tonabersat
- Placebo (Placebo Comparator): IFX-LC001Tonabersat tablets 40mg tablets or placebo Take two tablets once per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tonabersat — Tonabersat 40mg. Two tablets per day
  Other Names: Xiflam
  Arms: Experimental
Drug: Placebo — Placebo 40mg, Two tablets per day
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of Xiflam versus Placebo in patients who present with signs and symptoms of Long COVID.

Xiflam (n=10) or placebo (n=5) will be administered orally once a day (QD) for 12 weeks.

DETAILED DESCRIPTION:
This is a Phase 2a randomized, masked, placebo-controlled clinical trial to evaluate the safety and efficacy of Xiflam for use in patients with signs/symptoms of Long COVID. Patients will be randomized to Xiflam the study drug (n=10) or Placebo (n=5). Both Xiflam and Placebo will be taken once daily by mouth for 12 weeks.

I. Baseline Screening Visit After obtaining informed consent and before treatment is initiated, an initial study visit will be conducted in person to confirm subject eligibility. Subjects will be asked complete a baseline questionnaire to assess signs and symptom severity. During this screening visit, a baseline blood sample will be obtained to determine any changes over time in any of the measured parameters. These include biomarkers of inflammation. Additional study procedures occurring during the baseline/screening phase of this study are outlined in the protocol. Patients who are found not to meet inclusion criteria, will not be entered into the treatment Phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have tested positive for COVID-19 irrespective of variant or timeframe.
2. Developed signs and symptoms of the disease as described by the Centers for Disease Control and Prevention (CDC) and World Health Organization (WHO).
3. Have recovered from the infection (tested negative for COVID-19).
4. Following negative COVID-19 testing, continued to demonstrate signs/symptoms which were not pre-existing. The signs/symptoms must have persisted for 12 weeks or more.
5. Have had a persistent recurrence of a disease state (e.g., posterior uveitis, extreme fatigue etc.) that occurred following COVID-19 infection.
6. Female subjects must be:

   1. Women of non-child-bearing potential, or
   2. Women of child-bearing potential with a negative pregnancy test at screening, must agree to use approved methods of contraception for the duration of the study and refrain from breastfeeding for the duration of the study.
7. Males with female partners of child-bearing potential must agree to use approved methods of contraception and agree to refrain from donating sperm for the duration of the study.
8. Willing and able to give informed consent and to comply with the study procedures and assessments.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following exclusion criteria apply:

1. No proof of having tested positive for COVID-19 infection at any time.
2. Presence of an active ocular/systemic disease that in the opinion of the Investigator existed prior to COVID-19 infection and is not likely a LC related condition.
3. Intraocular surgery (including lens replacement surgery) within 3 months prior to randomization.
4. History of laser therapy in the macular region.
5. Any ocular or systemic condition that in the opinion of the Investigator is not LC related (e.g., pre-existing cataract) that may require surgery or medical intervention during the study period.
6. Participation in any systemic experimental treatment or any other systemic investigational new drug within 90 days prior to the start of study treatment.
7. Any screening laboratory value (hematology, serum chemistry or urinalysis) that in the opinion of the Investigator is clinically significant and not suitable for study participation.
8. Known hypersensitivity to Xiflam™ or excipients.
9. Known history of alcohol and/or drug abuse within 12 months prior to Visit 1 Screening that, in the opinion of the Investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 weeks
  Primary outcomes are change from baseline for signs and symptoms measured by a Visual Analogue Scale (VAS) instrument. Reporting done by the patient on a 0-100 scale. Scale measures severity from none (0) to severe (100) for multiple signs and symptoms, for the different systems involved in this disease state (see below)
  1. General health
  2. Neurological signs/symptoms
  3. Ocular signs/symptoms
  4. Respiratory signs/symptoms
  5. Gastrointestinal signs/symptoms
  6. Cardiovascular signs/symptoms
  7. Musculoskeletal signs/symptoms
  8. Dermatological signs/symptoms
  9. Mental Health signs/symptoms
  10. Miscellaneous signs/symptoms which may not be captured above.
  Since Long COVID is a multi-system disease, patients will only score on the severity scale of the signs/symptoms which are of clinical significance to that particular patient.

SECONDARY OUTCOMES:
Secondary Endpoint | 12 weeks
  Complete Blood Count (CBC) including biomarkers of inflammation Physical Examination including electrocardiogram (EKG)
  Change in laboratory values including inflammatory markers, e.g., C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), Antinuclear Antibody (ANA)

OTHER OUTCOMES:
Safety Endpoint | 12 weeks
  Incidence and severity of ocular and systemic treatment emergent adverse events (TEAE)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chang, MD, Principal Investigator — Massachusetts Eye Research and Surgery Institution (MERSI)
Locations (1):
- Massachusetts Eye Research and Surgery Institution (MERSI), Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No